CLINICAL TRIAL: NCT03901092
Title: A Reader Study to Assess Accuracy and Reliability of Flortaucipir F 18 PET Scan Interpretation
Brief Title: A Reader Study to Assess Accuracy and Reliability of Flortaucipir F 18 Positron Emission Tomography (PET) Scan Interpretation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-FR01
Record Dates: First submitted 2019-03-27; First posted 2019-04-03 (Actual); Results first posted 2020-08-11 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer Disease
Keywords: flortaucipir F 18; Positron Emission Tomography; 18F-AV-1451; Diagnostic imaging; Tau imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Intervention Model Description: Physician PET scan readers are participants, blinded to demographic and clinical data from the source PET scans.
Masking Description: PET scans were obtained in an open-label fashion.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Flortaucipir PET Scan (Experimental): Scans previously acquired from Study A16 (NCT02516046) and A05 (NCT02016560) will be read by independent, blinded readers.
  Interventions: Drug: flortaucipir F 18

INTERVENTIONS:
Drug: flortaucipir F 18 — No study drug will be administered.
  Other Names: 18F-AV-1451; [F-18]T807; LY3191748

SUMMARY:
This study will evaluate the performance of physician readers trained to read flortaucipir-PET (positron emission tomography) scans.

ELIGIBILITY:
Scan Reader Criteria (5 total):

* Board-certified in radiology or nuclear medicine
* Professional experience interpreting PET scans
* Naive to study protocol
* No previous training or exposure to Avid Flortaucipir F 18 read methodology

Scan Criteria:

- Previous enrollment in Study A05 confirmatory cohort (NCT02016560), or A16 (NCT02516046)

Scan Study Population Criteria for FR01 (A05 confirmatory cohort):

* Cognitively-impaired
* mild cognitive impairment (MCI) or dementia with suspected neurodegenerative cause
* mini-mental status exam (MMSE) score of 20-27, inclusive

Scan Study Population Criteria for FR01 (Study A16):

* Subjects at end of life (less than or equal to 6 months)
* Imaged with flortaucipir F18 and came to autopsy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Avid Radiopharmaceuticals
Locations (1):
- American College of Radiology, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were not recruited for this study. Study scans were selected from 2 previously completed imaging studies. Scans previously acquired from Study A16 (NCT02516046) and A05 (NCT02016560) were read by 5 independent, blinded to other study information.
Groups:
- All Autopsy Cases: Cases that had a valid scan and came to autopsy in in study A16 and the A16 supplemental cohort
- Non-Autopsy Cases: Mild cognitive impairment (MCI) and AD cases from the A05 confirmatory cohort
Period: Overall Study
Arm/Group | All Autopsy Cases | Non-Autopsy Cases
Started | 83 | 159
Completed | 83 | 159
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Cases: All eligible subject scans from contributing studies
Arm/Group | All Cases
Number analyzed (Participants) | 242
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline analysis includes Study A16 autopsy cases (n=83) and Study A05 Non-autopsy cases (n=159).
  years
    Study A16 Autopsy Cases: number analyzed (Participants) | 83
    Study A16 Autopsy Cases | 81.6 (9.91)
    Study A05 Non-autopsy Cases: number analyzed (Participants) | 159
    Study A05 Non-autopsy Cases | 72.9 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline analysis includes Study A16 autopsy cases (n=83) and Study A05 Non-autopsy cases (n=159).
  Participants
    Study A16 Autopsy Cases: number analyzed (Participants) | 83
    Study A16 Autopsy Cases: Female | 41
    Study A16 Autopsy Cases: Male | 42
    Study A05 Non-autopsy Cases: number analyzed (Participants) | 159
    Study A05 Non-autopsy Cases: Female | 74
    Study A05 Non-autopsy Cases: Male | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Baseline analysis includes Study A16 autopsy cases (n=83) and Study A05 Non-autopsy cases (n=159).
  Participants
    Study A16 Autopsy Cases: number analyzed (Participants) | 83
    Study A16 Autopsy Cases: Hispanic or Latino | 4
    Study A16 Autopsy Cases: Not Hispanic or Latino | 79
    Study A16 Autopsy Cases: Unknown or Not Reported | 0
    Study A05 Non-autopsy Cases: number analyzed (Participants) | 159
    Study A05 Non-autopsy Cases: Hispanic or Latino | 9
    Study A05 Non-autopsy Cases: Not Hispanic or Latino | 150
    Study A05 Non-autopsy Cases: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Baseline analysis includes Study A16 autopsy cases (n=83) and Study A05 Non-autopsy cases (n=159).
  Participants
    Study A16 Autopsy Cases: number analyzed (Participants) | 83
    Study A16 Autopsy Cases: American Indian or Alaska Native | 0
    Study A16 Autopsy Cases: Asian | 1
    Study A16 Autopsy Cases: Native Hawaiian or Other Pacific Islander | 0
    Study A16 Autopsy Cases: Black or African American | 1
    Study A16 Autopsy Cases: White | 81
    Study A16 Autopsy Cases: More than one race | 0
    Study A16 Autopsy Cases: Unknown or Not Reported | 0
    Study A05 Non-autopsy Cases: number analyzed (Participants) | 159
    Study A05 Non-autopsy Cases: American Indian or Alaska Native | 0
    Study A05 Non-autopsy Cases: Asian | 2
    Study A05 Non-autopsy Cases: Native Hawaiian or Other Pacific Islander | 0
    Study A05 Non-autopsy Cases: Black or African American | 3
    Study A05 Non-autopsy Cases: White | 154
    Study A05 Non-autopsy Cases: More than one race | 0
    Study A05 Non-autopsy Cases: Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Objective 1 Analysis 1: Diagnostic Performance of Individual Readers (NFT Score)
Description: Sensitivity and specificity of 5 independent readers' interpretations of ante-mortem 18F-AV-1451 PET imaging for detection of a pattern of 18F-AV-1451 neocortical uptake that corresponds to neurofibrillary tangles (NFT) Score of B3 (Hyman et al., 2012; Montine et al., 2012). NFT B scores range from B0 (no NFTs in the brain) to B3 (widespread NFTs in the brain). Sensitivity and specificity are percentages that can range from 0 to 100%. The hypothesis tested was that, of the 5 independent imaging physicians, at least 3 will have the lower bounds of 2-sided 95% CIs ≥50%, for both sensitivity and specificity.
Time Frame: baseline scan
Population: Analysis included all autopsy subjects with an evaluable flortaucipir PET scan interpretation (n=82). One autopsy subject scan was rated as unevaluable. n=47 were truth positive for NFTs. n=35 were truth negative for NFTs.
Measure: Number (95% Confidence Interval); unit: percentage of cases correctly identified
Groups:
- Sensitivity of Flortaucipir vs Autopsy NFT Score: Subjects with a positive autopsy NFT score truth standard (NFT B3)
- Specificity of Flortaucipir vs Autopsy NFT Score: Subjects with a negative autopsy NFT score truth standard (NFT B2 or lower)
Arm/Group | Sensitivity of Flortaucipir vs Autopsy NFT Score | Specificity of Flortaucipir vs Autopsy NFT Score
Number analyzed (Participants) | 47 | 35
percentage of cases correctly identified
  Reader 1 | 91.5 [80.07 to 96.64] | 77.1 [60.98 to 87.93]
  Reader 2 | 89.4 [77.41 to 95.37] | 91.4 [77.62 to 97.04]
  Reader 3 | 87.2 [74.83 to 94.02] | 85.7 [70.62 to 93.74]
  Reader 4 | 93.6 [82.84 to 97.81] | 62.9 [46.34 to 76.83]
  Reader 5 | 89.4 [77.41 to 95.37] | 77.1 [60.98 to 87.93]

2. Primary Outcome: Primary Objective 1 Analysis 2: Diagnostic Performance of Individual Readers (NIA-AA Autopsy Diagnosis)
Description: Sensitivity and specificity of 5 independent readers' interpretations of ante-mortem 18F-AV-1451 PET imaging for detection of a pattern of 18F-AV-1451 neocortical uptake that corresponds to high levels of AD neuropathologic change (High ADNC) as defined by National Institute on Aging-Alzheimer's Association (NIA-AA) criteria (see Hyman et al. 2012). ADNC categories are None, Low, Intermediate and High, with High indicating the most severe level of AD-related pathology changes in the brain. The hypothesis tested was that, of the 5 independent imaging physicians, at least 3 will have the lower bounds of 2-sided 95% CIs ≥50%, for both sensitivity and specificity.
Time Frame: baseline scan
Population: Analysis included all autopsy subjects with an evaluable flortaucipir PET scan interpretation (n=82). One autopsy subject scan was rated as unevaluable. n=41 were truth positive. n=41 were truth negative.
Measure: Number (95% Confidence Interval); unit: percentage of cases correctly identified
Groups:
- Sensitivity of Flortaucipir vs NIA-AA Autopsy Diagnosis: Subjects with a positive truth standard (High ADNC)
- Specificity of Flortaucipir vs NIA-AA Autopsy Diagnosis: Subjects with a negative truth standard (No/Low/Intermediate ADNC)
Arm/Group | Sensitivity of Flortaucipir vs NIA-AA Autopsy Diagnosis | Specificity of Flortaucipir vs NIA-AA Autopsy Diagnosis
Number analyzed (Participants) | 41 | 41
percentage of cases correctly identified
  Reader 1 | 95.1 [83.86 to 98.65] | 70.7 [55.52 to 82.39]
  Reader 2 | 95.1 [83.86 to 98.65] | 85.4 [71.56 to 93.12]
  Reader 3 | 95.1 [83.86 to 98.65] | 82.9 [68.74 to 91.47]
  Reader 4 | 97.6 [87.40 to 99.57] | 58.5 [43.37 to 72.24]
  Reader 5 | 95.1 [83.86 to 98.65] | 73.2 [58.07 to 84.31]

3. Primary Outcome: Primary Objective 2: Inter-reader Reliability of Reader Interpretation of Flortaucipir-PET Imaging
Description: As measured by Fleiss' Kappa across all scans read. Fleiss' kappa is a statistical measure for assessing the reliability of agreement between a fixed number of raters when assigning categorical ratings to a number of items or classifying items. Fleiss' kappa can range from 0 to 1 with 1 indicating perfect agreement between the readers. Scan results binarized as positive AD pattern versus negative AD pattern. Results are displayed as percentage of agreement for individual reader pairs, computed as follows: number of images for which reader had the same interpretation divided by the total number of images evaluated, multiplied by 100%.
Time Frame: baseline scan
Population: Analysis included all subjects who had a valid flortaucipir PET scan in the autopsy and non-autopsy groups (n=241)
Measure: Number; unit: percentage agreement of cases
Groups:
- All Cases: All autopsy and non-autopsy cases
Arm/Group | All Cases
Number analyzed (Participants) | 241
percentage agreement of cases
  Reader 1 v Reader 2 | 95.0
  Reader 1 v Reader 3 | 93.4
  Reader 1 v Reader 4 | 94.6
  Reader 1 v Reader 5 | 97.1
  Reader 2 v Reader 3 | 97.1
  Reader 2 v Reader 4 | 91.3
  Reader 2 v Reader 5 | 94.6
  Reader 3 v Reader 4 | 91.3
  Reader 3 v Reader 5 | 93.8
  Reader 4 v Reader 5 | 95.0
Statistical Analysis 1: Comparison: All Cases; Fleiss' kappa is a statistical measure for assessing the reliability of agreement between a fixed number of raters when assigning categorical ratings to a number of items or classifying items. The primary hypothesis to be tested was that the lower bound of two-sided 95% confidence interval of Fleiss' Kappa will be greater than or equal to 0.6; Test type: Other; Fleiss' kappa = 0.87, 95% CI 2-sided [0.83 to 0.91]

4. Secondary Outcome: Secondary Objective 1 Analysis 1: Diagnostic Performance of τAD++ Flortaucipir PET Images to Detect B3 NFTs
Description: Flortaucipir F 18 PET imaging will be classified by each reader as either neocortical uptake not consistent with AD (τAD-), neocortical uptake consistent with AD (τAD+), or neocortical uptake consistent with AD with uptake beyond the temporal/occipital regions (τAD++). NFT scoring is according to Hyman, et al 2012. Truth positive is a NFT B3 score. Truth negative is NFT <B3 score.
Time Frame: baseline scan
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage cases correctly identified
Groups:
- Sensitivity of Flortaucipir tAD++ vs Autopsy NFT Score: Subjects with a positive autopsy NFT score truth standard (NFT B3)
- Specificity of Flortaucipir tAD++ vs Autopsy NFT Score: Subjects with a negative autopsy NFT score truth standard (NFT B2 or lower)
Arm/Group | Sensitivity of Flortaucipir tAD++ vs Autopsy NFT Score | Specificity of Flortaucipir tAD++ vs Autopsy NFT Score
Number analyzed (Participants) | 47 | 35
percentage cases correctly identified
  Reader 1 | 87.2 [74.83 to 94.02] | 88.6 [74.05 to 95.46]
  Reader 2 | 80.9 [67.46 to 89.58] | 100.0 [90.11 to 100.00]
  Reader 3 | 76.6 [62.78 to 86.40] | 94.3 [81.39 to 98.42]
  Reader 4 | 89.4 [77.41 to 95.37] | 82.9 [67.32 to 91.90]
  Reader 5 | 83.0 [69.86 to 91.11] | 94.3 [81.39 to 98.42]

5. Secondary Outcome: Secondary Objective 1 Analysis 2: Diagnostic Performance of τAD++ Flortaucipir PET Images to Detect High ADNC
Description: Sensitivity and specificity of 5 independent readers' interpretations of ante-mortem 18F-AV-1451 PET imaging for detection of a pattern of 18F-AV-1451 neocortical uptake that corresponds to high levels of AD neuropathologic change (High ADNC) as defined by National Institute on Aging-Alzheimer's Association (NIA-AA) criteria (Hyman et al. 2012). Truth positive is a High ADNC score. Truth negative is No/Low/Intermediate ADNC score.
Time Frame: baseline scan
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of cases correctly identified
Groups:
- Sensitivity: Sensitivity individual Flortaucipir PET scan interpreted as τAD++ pattern versus NIA-AA autopsy Diagnosis Truth Standard
- Specificity: Specificity individual Flortaucipir PET scan interpreted as τAD++ pattern versus NIA-AA autopsy Diagnosis Truth Standard
Arm/Group | Sensitivity | Specificity
Number analyzed (Participants) | 41 | 41
percentage of cases correctly identified
  Reader 1 | 92.7 [80.57 to 97.48] | 82.9 [68.74 to 91.47]
  Reader 2 | 85.4 [71.56 to 93.12] | 92.7 [80.57 to 97.48]
  Reader 3 | 85.4 [71.56 to 93.12] | 92.7 [80.57 to 97.48]
  Reader 4 | 92.7 [80.57 to 97.48] | 75.6 [60.66 to 86.17]
  Reader 5 | 87.8 [74.46 to 94.68] | 87.8 [74.46 to 94.68]

6. Secondary Outcome: Secondary Objective 2: Inter-reader Reliability of Reader Interpretation of τAD++ Flortaucipir PET Images
Description: Overall reader agreement as measured by Fleiss' Kappa statistic. Scan results binarized as τAD++ versus τAD+/τAD-. Results are displayed as percentage of agreement for individual reader pairs, computed as follows: number of images for which reader had the same interpretation divided by the total number of images evaluated, multiplied by 100%.
Time Frame: baseline scan
Population: Analysis included all subjects who had a valid flortaucipir PET scan in the autopsy and non-autopsy groups (n=241)
Measure: Number; unit: percentage agreement of cases
Arm/Group | All Cases
Number analyzed (Participants) | 241
percentage agreement of cases
  Reader 1 v Reader 2 | 92.5
  Reader 1 v Reader 3 | 90.0
  Reader 1 v Reader 4 | 91.3
  Reader 1 v Reader 5 | 95.0
  Reader 2 v Reader 3 | 91.7
  Reader 2 v Reader 4 | 90.5
  Reader 2 v Reader 5 | 94.2
  Reader 3 v Reader 4 | 88.8
  Reader 3 v Reader 5 | 92.5
  Reader 4 v Reader 5 | 92.9
Statistical Analysis 1: Comparison: All Cases; [analysis description as in outcome 3, analysis 1]; Test type: Other; Fleiss' kappa = 0.84, 95% CI 2-sided [0.80 to 0.88]

7. Secondary Outcome: Secondary Objective 3: Inter-reader Reliability of Flortaucipir PET Scan Interpretation in the Population of Intended Use
Description: Reader agreement measured by Fleiss' Kappa across scans from non-autopsy cases from Study A05. Scan results binarized as positive for AD pattern versus negative for AD pattern. Results are displayed as percentage of agreement for individual reader pairs, computed as follows: number of images for which reader had the same interpretation divided by the total number of images evaluated, multiplied by 100%.
Time Frame: baseline scan
Population: Non-autopsy cases from Study A05
Measure: Number; unit: percentage agreement of cases
Groups:
- A05 Cases: All non-autopsy cases from the Study A05 population of intended use
Arm/Group | A05 Cases
Number analyzed (Participants) | 159
percentage agreement of cases
  Reader 1 v Reader 2 | 97.5
  Reader 1 v Reader 3 | 93.1
  Reader 1 v Reader 4 | 95.6
  Reader 1 v Reader 5 | 97.5
  Reader 2 v Reader 3 | 93.1
  Reader 2 v Reader 4 | 94.3
  Reader 2 v Reader 5 | 96.2
  Reader 3 v Reader 4 | 93.7
  Reader 3 v Reader 5 | 93.1
  Reader 4 v Reader 5 | 96.9
Statistical Analysis 1: Comparison: A05 Cases; Fleiss' kappa is a statistical measure for assessing the reliability of agreement between a fixed number of raters when assigning categorical ratings to a number of items or classifying items. The hypothesis to be tested was that the lower bound of two-sided 95% confidence interval of Fleiss' Kappa will be greater than or equal to 0.6; Test type: Other; Fleiss' kappa = 0.90, 95% CI 2-sided [0.85 to 0.95]

8. Secondary Outcome: Secondary Objective 4: Intra-reader Reliability of Reader Interpretation of Flortaucipir-PET Imaging
Description: Cohen's Kappa will be calculated for each of 5 readers to assess the intra-reader reliability of flortaucipir F 18 PET scan visual interpretation. The statistic takes into account the possibility of the agreement occurring by chance. Cohen's kappa values range from 0 to 1 with 1 representing perfect agreement. Results are displayed as percentage of agreement within a reader, computed as follows: number of images for which reader had the same interpretation at initial and second read divided by the total number of images evaluated twice by a reader, multiplied by 100%.
Time Frame: baseline scan
Population: 20 scans read twice to assess the intra-reader reliability
Measure: Number; unit: percentage agreement of cases
Groups:
- Randomly Selected Re-reads: Cases randomly selected to be read twice by the same reader
Arm/Group | Randomly Selected Re-reads
Number analyzed (Participants) | 20
percentage agreement of cases
  Reader 1 | 95.0
  Reader 2 | 85.0
  Reader 3 | 80.0
  Reader 4 | 95.0
  Reader 5 | 90.0
Statistical Analysis 1: Comparison: Randomly Selected Re-reads; Cohen's kappa statistic for Reader 1; Test type: Other; Cohen's kappa = 0.89, 95% CI 2-sided [0.69 to 1.00]
Statistical Analysis 2: Comparison: Randomly Selected Re-reads; Cohen's kappa statistic for Reader 2; Test type: Other; Cohen's kappa = 0.71, 95% CI 2-sided [0.41 to 1.00]
Statistical Analysis 3: Comparison: Randomly Selected Re-reads; Cohen's kappa statistic for Reader 3; Test type: Other; Cohen's kappa = 0.60, 95% CI 2-sided [0.24 to 0.95]
Statistical Analysis 4: Comparison: Randomly Selected Re-reads; Cohen's kappa statistic for Reader 4; Test type: Other; Cohen's kappa = 0.89, 95% CI 2-sided [0.67 to 1.00]
Statistical Analysis 5: Comparison: Randomly Selected Re-reads; Cohen's kappa statistic for Reader 5; Test type: Other; Cohen's kappa = 0.79, 95% CI 2-sided [0.52 to 1.00]

ADVERSE EVENTS:
Time Frame: Not applicable. Adverse events were not assessed during this study.
Description: Adverse events were not assessed during this study.
Groups:
- All Cases: No study drug will be administered. Scans previously acquired from Study A16 (NCT02516046) and A05 (NCT02016560) will be read by independent, blinded readers.
Arm/Group | All Cases
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03901092/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT03901092/SAP_001.pdf